CLINICAL TRIAL: NCT05465551
Title: Development of a Dyadic Stress Management Toolkit for People Living With Dementia and Their Care Partners
Brief Title: Stress Management Toolkit for People Living With Dementia and Their Care Partners
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00110944; P30AG072958 (NIH)
Record Dates: First submitted 2022-06-27; First posted 2022-07-20 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Dementia; Stress; Caregiver Burden
Keywords: Nonpharmacological interventions
MeSH Terms: conditions — Dementia; Caregiver Burden

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stress Management Toolkit Prototype Development (No Intervention): 3-4 qualitative focus groups (n=3-4 dyads/group) will be held to explore experiences, perceptions, preferences, and recommendations of dementia-caring dyads regarding stress, stress management, and key components and features of a stress management toolkit. Eligible tools for the toolkit include low burden, high safety tools (e.g., weighted blankets, robotic pets and baby dolls, guided journals, aromatherapy, bright light therapy devices, massage and acupressure tools).
- Stress Management Toolkit Prototype User Testing (Experimental): 10 dyads will use the toolkit for 2 weeks in their own homes. Feedback on usability, feasibility, and acceptability will be collected through questionnaires and focus groups. Stress-related, participant-reported outcomes (e.g., neuropsychiatric symptoms of dementia, caregiver stress, dyadic relationship strain), and salivary cortisol biospecimens will be collected at baseline and end of week 2, to explore their utility as endpoints in a future pilot study to examine efficacy.
  Interventions: Combination Product: Stress Management Toolkit

INTERVENTIONS:
Combination Product: Stress Management Toolkit — The toolkit will be a home-based, dyadic tangible toolkit comprised of simple tools to help people living with dementia (PLWD) and their care partners manage stress at home. Potential tools for the toolkit includes low burden, high safety tools such as weighted blankets, robotic pets and baby dolls, guided journals, aromatherapy and bright light therapy devices, and massage and acupressure tools. The tookit will also include user-safety guidelines and directions on how to use each tool. Tools will be included for participants with dementia and care partners.
  Arms: Stress Management Toolkit Prototype User Testing

SUMMARY:
The purpose of this study is to develop a prototype of a home-based, dyadic tangible toolkit comprised of simple tools to help people living with dementia (PLWD) and their care partners manage stress at home.

A human-centered design approach will be used to develop and user-test a prototype of a dyadic, tangible stress-management toolkit with and for PLWD and their care partners; and to explore the feasibility of collecting several stress-related outcomes. A total of 4 focus groups (n=3-4 dyads/group) will be convened to explore the experiences, perceptions, preferences, and recommendations of dementia-caring dyads regarding stress, stress management, and key components and features of a stress management toolkit. Eligible tools for the toolkit include low burden, high safety tools such as weighted blankets, robotic pets and baby dolls, guided journals, aromatherapy and bright light therapy devices, and massage and acupressure tools. Ten dyads who were not involved in prototype development will then use the toolkit for 2 weeks. Feedback on usability, feasibility, and acceptability will be collected through questionnaires (end of weeks 1 and 2) and 3 focus groups (3-4 dyads/group at end of week 2). We will collect stress-related, participant-reported outcomes (e.g., neuropsychiatric symptoms of dementia, caregiver stress, dyadic relationship strain), and saliva biospecimens from participants with dementia and their care partners at baseline and end of week 2, to explore their utility as endpoints in a future toolkit intervention that uses a single-arm, pre-post study design. Results will yield valuable data to support development and preliminary testing of a stress management toolkit intervention in a future pilot study.

This study involves human subjects and is expected to yield no more than minimal risk. Tools eligible for the toolkit must have demonstrated high degrees of safety in prior research. Major risks for participation include the potential for negative emotional responses to focus group discussions and surveys pertaining to stress, excess time burden to participate in the study, and breach of confidentiality. It is not anticipated, but there is a potential for physical discomfort if tools are not used as directed, which is why the toolkits will include a user guide outlining safety information, which a research team member will review with each participant prior to use.

ELIGIBILITY:
Inclusion criteria for participants with dementia are:

* age 60 years and over with a diagnosis of dementia of any type
* able to express self verbally
* English speaking.

Exclusion criteria for participants with dementia is:

• has a hearing or visual impairment that limits their ability to participate in the screening process or to participate in a focus group.

Inclusion criteria for care partner participants are:

* age 21 years and older
* identify as a primary care partner of someone with dementia
* English speaking

Exclusion criteria for care partner participants is:

• has a hearing or visual impairment that limits their ability to participate in the screening process or to participate in a focus group.

Dyadic eligibility criteria include:

* both the PLWD and care partner reside in the same household or personal residence in the community
* dyad has lived together for at least 1 month
* dyad has telephone or internet access
* Dyads will be excluded if they reside in assisted living or other long-term care setting.

Dyads participating in user-testing phase will also be excluded if either member:

* currently receives cytokine-based therapy
* currently receives radiation therapy to the salivary glands or thyroid
* are diagnosed with Cushing or Addison's disease

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2022-12-20 (Actual); Primary Completion 2025-01-06 (Actual); Study Completion 2025-01-06 (Actual)

PRIMARY OUTCOMES:
Frequency of toolkit use | End of week 1 of user-testing period
  Number of days toolkit was used over the last week (range 0-7) will be assessed among participants enrolled in user-testing arm.
Frequency of toolkit use | End of week 2 of user-testing period
  Number of days toolkit was used over the last week (range 0-7) will be assessed among participants enrolled in user-testing arm.
Enrollment rate | Through study completion, an average of 1 year
  Percentage of participant dyads enrolled/dyads screened in user-testing arm.
Withdrawal rate | Through study completion, an average of 1 year
  Percentage of dyads that withdraw/dyads enrolled in user-testing arm.
Frequency of adverse events and injuries | Through study completion, an average of 1 year
  Number of adverse events and injuries reported in user-testing arm.
Participant satisfaction with toolkit, as assessed using a toolkit satisfaction scale | Within 1 week after user-testing period
  Investigator developed multi-item satisfaction scale will include Likert-scaled items pertaining to satisfaction with design and delivery of the toolkit among participants in the user-testing arm; item ranges 1=not satisfied at all to 5 very satisfied). Scores will be averaged to yield and overall satisfaction score with higher scores indicating a greater degree of satisfaction.
Participant perceived benefit with toolkit, as assessed using a toolkit benefit scale | Within 1 week after user-testing period
  Investigator developed multi-item benefit scale will include Likert-scaled items pertaining to perceived benefit from the toolkit among participants in the user-testing arm; item ranges 1=not beneficial at all to 5 very beneficial). Scores will be averaged to yield and overall benefit score with higher scores indicating a greater degree of benefit.

SECONDARY OUTCOMES:
Percentage of participant completion of neuropsychiatric symptoms of dementia outcome measure, as assessed using the Neuropsychiatric Inventory-Questionnaire | Baseline, pre user-testing period
  Percentage of participant completion for this measure will be calculated for participants enrolled in the user-testing arm (Number of participants who complete the measure at baseline/total number of participants enrolled in user-testing arm). NPI assesses severity (1=mild, 2=moderate, 3=severe) and caregiver distress (range 0=not distressing at all to 5 extreme or very severe) of 12 domains of neuropsychiatric symptoms of dementia. Higher scores indicate more severe or distressing symptoms.
Percentage of participant completion of neuropsychiatric symptoms of dementia outcome measure, as assessed using the Neuropsychiatric Inventory-Questionnaire | Within 1 week after user-testing period
  Percentage of participant completion for this measure will be calculated for participants enrolled in the user-testing arm (Number of participants who complete the measure at post user-testing/total number of participants enrolled in user-testing arm). NPI assesses severity (1=mild, 2=moderate, 3=severe) and caregiver distress (range 0=not distressing at all to 5 extreme or very severe) of 12 domains of neuropsychiatric symptoms of dementia. Higher scores indicate more severe or distressing symptoms.
Percentage of participant completion of caregiver stress outcome measure, as assessed using the Perceived Stress Scale | Baseline, pre user-testing period
  Percentage of participant completion for this measure will be calculated for participants enrolled in the user-testing arm (Number of participants who complete the measure at baseline/total number of participants enrolled in user-testing arm). The Perceived Stress Scale is a 10-item measure that assesses recent stress-related thoughts and feelings on 5-point scale with higher scores indicating higher levels of stress.
Percentage of participant completion of caregiver stress outcome measure, as assessed using the Perceived Stress Scale | Within 1 week after user-testing period
  Percentage of participant completion for this measure will be calculated for participants enrolled in the user-testing arm (Number of participants who complete the measure at post user-testing/total number of participants enrolled in user-testing arm). The Perceived Stress Scale is a 10-item measure that assesses recent stress-related thoughts and feelings on 5-point scale with higher scores indicating higher levels of stress.
Percentage of participant completion of dyadic relationship strain outcome measure, as assessed using the Dyadic Relationship Scale | Baseline, pre user-testing period
  Percentage of participant completion for this measure will be calculated for participants enrolled in the user-testing arm (Number of participants who complete the measure at baseline/total number of participants enrolled in user-testing arm). The Dyadic Relationship Scale includes a care recipient 10-item version and care partner specific 11-item version. Both scales measure dyadic strain and positive dyadic interaction. Total scores range from 0-30 for the care recipient version, and 0-33 for care partner specific, with higher scores indicative of higher levels of dyadic strain.
Percentage of participant completion of dyadic relationship strain outcome measure, as assessed using the Dyadic Relationship Scale | Within 1 week after user-testing period
  Percentage of participant completion for this measure will be calculated for participants enrolled in the user-testing arm (Number of participants who complete the measure at post user-testing/total number of participants enrolled in user-testing arm). The Dyadic Relationship Scale includes a care recipient 10-item version and care partner specific 11-item version. Both scales measure dyadic strain and positive dyadic interaction. Total scores range from 0-30 for the care recipient version, and 0-33 for care partner specific, with higher scores indicative of higher levels of dyadic strain.
Percentage of participant completion of physiologic stress outcome measure, as assessed through salivary cortisol biospecimens | Baseline, pre user-testing period
  Percentage of participant completion for this measure will be calculated for participants enrolled in the user-testing arm (Total number of biospecimen samples collected among participants at baseline/total number of participants enrolled in user-testing arm*5).
  Salivary cortisol biospecimens will be collected using salivary sample kits sent to participants' homes by mail. Participants with dementia and care partners will each be asked to collect 5 samples at baseline and will collect samples themselves in their own homes with guidance and support from research team. Samples will be mailed back to research team using preaddressed, prestamped envelopes.
Percentage of participant completion of physiologic stress outcome measure, as assessed through salivary cortisol biospecimens | Within 1 week after user-testing period
  Percentage of participant completion for this measure will be calculated for participants enrolled in the user-testing arm (Total number of biospecimen samples collected among participants at post user-testing/total number of participants enrolled in user-testing arm*5).
  Salivary cortisol biospecimens will be collected using salivary sample kits sent to participants' homes by mail. Participants with dementia and care partners will each be asked to collect 5 samples at post user-testing and will collect samples themselves in their own homes with guidance and support from research team. Samples will be mailed back to research team using preaddressed, prestamped envelopes.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa L Harris, PhD, Principal Investigator — Duke University School of Nursing; Susan N Hastings, MD, Principal Investigator — Duke University
Locations (1):
- Caregiver and dementia community support organizations, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Harris M, Van Houtven C, Hastings S. Development of a Home-Based Stress Management Toolkit for Dementia Caring Dyads: Protocol for a Pilot Intervention Development and Feasibility Study. JMIR Res Protoc. 2022 Dec 14;11(12):e43098. doi: 10.2196/43098. PMID 36399169